CLINICAL TRIAL: NCT03049618
Title: A Phase IIa Trial of sEphB4-HSA in Combination With Anti PD-1 Antibody (Pembrolizumab, MK3475) in Patients With Non-small Cell Lung and Head/Neck Cancer
Brief Title: Recombinant EphB4-HSA Fusion Protein and Pembrolizumab, MK-3475
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0S-16-8; NCI-2017-00189 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-16-8 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: ALK Gene Mutation; BRAF Gene Mutation; EGFR Gene Mutation; Head and Neck Squamous Cell Carcinoma; Metastatic Head and Neck Carcinoma; Recurrent Head and Neck Carcinoma; Recurrent Non-Small Cell Lung Carcinoma; ROS1 Gene Mutation; Stage III Non-Small Cell Lung Cancer; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Head and Neck Cancer Cohort (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and recombinant EphB4-HSA fusion protein IV over 30 minutes on days 1, 8, and 15. Courses repeat every 3 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Biological: Recombinant EphB4-HSA Fusion Protein
- Non-Small Cell Lung Cancer Cohort (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and recombinant EphB4-HSA fusion protein IV over 30 minutes on days 1, 8, and 15. Courses repeat every 3 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Biological: Recombinant EphB4-HSA Fusion Protein

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Biological: Recombinant EphB4-HSA Fusion Protein — Given IV
  Other Names: sEphB4-HSA

SUMMARY:
This phase IIa trial studies how well recombinant EphB4-HSA fusion protein and pembrolizumab work in treating patients with non-small cell lung cancer that has spread to other places in the body or head and neck squamous cell cancer that has come back or spread to other places in the body. Recombinant EphB4-HSA fusion protein may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of cancer cells to grow and spread. Giving recombinant EphB4-HSA fusion protein and pembrolizumab may work better in treating patients with non-small cell lung or head and neck squamous cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate of the combination of pembrolizumab and recombinant EphB4-HSA fusion protein (sEphB4-HSA) as combination therapy.

SECONDARY OBJECTIVES:

I. Determine the biomarkers of response. II. Determine the unique toxicities of the combination of pembrolizumab and sEphB4-HSA.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and recombinant EphB4-HSA fusion protein IV over 30 minutes on days 1, 8, and 15. Courses repeat every 3 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* One of the following:

  * Locally advanced or metastatic non-small cell lung cancer that has progressed after at least 1 line of platinum based chemotherapy

    * Patients may have received up to 2 prior lines of chemotherapy
    * Patients with actionable alterations in EGFR/ALK/ROS1/BRAF must also have progressed after treatment with a tyrosine kinase inhibitor appropriate for their genetic alteration
    * Untreated patients who refuse 1st line platinum based chemotherapy are also eligible
  * Squamous cell carcinoma of the head and neck whose disease has progressed after at least 1 line of platinum based chemotherapy

    * Patients may have received up to 2 prior lines of chemotherapy
    * Untreated patients who refuse 1st line platinum based chemotherapy are also eligible
    * Patients who relapse within 6 months of adjuvant cisplatin based concurrent chemoradiation, or neoadjuvant cisplatin based therapy can be considered eligible without an additional course of platinum chemotherapy for relapsed disease
    * Patients may have either locally recurrent or distant metastatic disease
* Be willing and able to provide written informed consent/assent for the trial
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion after 2 cycles of therapy
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500 /mcL
* Platelets >= 100,000 / mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN
* Serum total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN OR =< 5 x ULN for subjects with liver metastases
* Albumin >= 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication

  * Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy

  * Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability; known brain metastases are considered active, if any of the following criteria is applicable:

  * Brain imaging during screening demonstrates progression of existing metastases and/or appearance of new lesions compared to brain imaging performed at least 4 weeks earlier
  * Neurological symptoms attributed to brain metastases have not returned to baseline
  * Steroids were used for brain metastases within 28 days of randomization
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Nieva, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study opened in March 2017 and closed in March 2021. All subjects were seen and treated in the medical clinics at the University of Southern California
Period: Overall Study
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Started | 25 | 17
Completed | 23 | 15
Not Completed | 2 | 2
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 1 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled patients are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort | Total
Number analyzed (Participants) | 25 | 17 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 10 | 4 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 20 | 8 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 19 | 13 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 17 | 8 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 17 | 42
Smoking Status [Count of Participants; unit: Participants]
  Never Smoke | 12 | 9 | 21
  Former Smoker | 11 | 7 | 18
  Current Smoker | 2 | 0 | 2
  Unknown | 0 | 1 | 1
ECOG Performance Status (PS) [Count of Participants; unit: Participants]
  Status 0 (Fully active without restriction) | 12 | 6 | 18
  Status 1 (Physically restricted but ambulatory and able to carry out light work) | 13 | 11 | 24
Site of Disease [Count of Participants; unit: Participants]
  Larynx | 4 | 0 | 4
  Lip and Oral Cavity | 14 | 0 | 14
  Nasal Cavity and Paranasal Sinuses | 5 | 0 | 5
  Pharynx | 2 | 0 | 2
  Lung - Bronchi, NOS | 0 | 10 | 10
  Lung - Lower Lobe | 0 | 4 | 4
  Lung - Middle Lobe | 0 | 1 | 1
  Lung - Upper Lobe | 0 | 2 | 2
Received Prior Surgery [Count of Participants; unit: Participants]
  Yes | 11 | 5 | 16
  No | 14 | 12 | 26
Received Prior Radiotherapy [Count of Participants; unit: Participants]
  Yes | 17 | 9 | 26
  No | 8 | 8 | 16
Received Prior Chemotherapy [Count of Participants; unit: Participants]
  Yes | 20 | 16 | 36
  No | 5 | 1 | 6
Number of Prior Regimens Received [Count of Participants; unit: Participants]
  0 | 5 | 1 | 6
  1 | 18 | 10 | 28
  2 | 2 | 5 | 7
  3 | 0 | 1 | 1
HPV Status [Count of Participants; unit: Participants] — Population: Enrollment to lung cohort terminated early so no specimen was processed
  Participants
    Negative: number analyzed (Participants) | 25 | 0 | 25
    Negative | 15 | 0 | 15
    Positive: number analyzed (Participants) | 25 | 0 | 25
    Positive | 10 | 0 | 10
P16 Gene Status [Count of Participants; unit: Participants] — Population: Enrollment to lung cohort terminated early so no specimen was processed
  Participants
    Negative: number analyzed (Participants) | 25 | 0 | 25
    Negative | 15 |  | 15
    Positive: number analyzed (Participants) | 25 | 0 | 25
    Positive | 10 |  | 10
EphrinB2 Status [Count of Participants; unit: Participants] — Population: Enrollment to lung cohort terminated early so no specimen was processed
  Participants
    Negative: number analyzed (Participants) | 25 | 0 | 25
    Negative | 9 | 0 | 9
    Positive: number analyzed (Participants) | 25 | 0 | 25
    Positive | 16 | 0 | 16
PDL-1 Status [Count of Participants; unit: Participants] — Population: Enrollment to lung cohort terminated early so no specimen was processed
  Participants
    Negative: number analyzed (Participants) | 25 | 0 | 25
    Negative | 13 | 0 | 13
    Positive: number analyzed (Participants) | 25 | 0 | 25
    Positive | 12 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Calculated based on the evaluable population of patients who received at least 1 dose of therapy. Overall response rate (ORR) is complete response (CR) + partial response (PR) recorded from study entry until disease progression based on RECIST v1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Up to 22 months
Population: Evaluable population of patients who received at least 1 dose of therapy. No statistical analysis is performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 17
Participants | 6 | 3

2. Secondary Outcome: Duration of Response
Description: Duration of response is measured from date of first confirmed response until date of disease progression.
Time Frame: Up to 22 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 6 | 17
Months | 3.7 [1.8 to 8.9] | 7.6 [1.6 to 28.0]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: The adverse events were graded as per common terminology criteria for adverse events(CTCAE) version 4.0. For a detailed list of adverse events refer to the adverse event module.
Time Frame: Adverse events were collected from first dose of study treatment up to 30 days after last dose of treatment, up to 21 months (number of treatment given ranged from 1 cycle to 30 cycles).
Population: All enrolled patients are included. No statistical analysis is performed.
Measure: Number; unit: participants
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 17
participants
  CTCAE grade 1 or 2 | 25 | 17
  CTCAE grade 3 or 4 | 23 | 17

4. Secondary Outcome: Overall Survival (OS)
Description: OS is the duration from study entry to death. Participants last known to be alive are censored at date of last contact.
Time Frame: Up to 41 months
Population: All enrolled patients are included. Statistical analysis was not performed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 17
Months | 8.6 [3.2 to 13.7] | 11.8 [4.2 to 30.1]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as duration of time from the first dose of study drug to the first documentation of Progressive Disease (PD) by investigator assessment using RECIST 1.1 or death on study due to any cause on or before the data cutoff date, whichever occurred first. PD: >=20% increase (>=5 mm absolute increase) in the sum of target lesion measurements, compared to the smallest sum on study (including baseline), or unequivocal progression of non-target lesions, evaluated as a whole, such that it is clear that treatment has failed, and disease is progressing, regardless of the status of the target lesions.
Time Frame: Up to 23 months
Population: All patients were included in the analysis. Statistical analysis was not performed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 17
Months | 2.6 [1.3 to 4.1] | 3.0 [1.2 to 6.1]

6. Other Pre Specified Outcome: Association of Biomarker With Overall Response Rate - HPV Status
Description: Overall response rate (ORR) is complete response (CR) + partial response (PR) recorded from study entry until disease progression based on RECIST v1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Up to 22 months
Population: Only the Head and Neck cancer cohort is being reported. No specimens were collected for the non-small cell lung cancer cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 0
Participants
  HPV Negative who achieved CR/PR: number analyzed (Participants) | 15 | 0
  HPV Negative who achieved CR/PR | 5 |
  HPV Positive who achieved CR/PR: number analyzed (Participants) | 10 | 0
  HPV Positive who achieved CR/PR | 1 |
Statistical Analysis 1: Comparison: Head and Neck Cancer Cohort; Test type: Other; p = 0.34, Fisher Exact

7. Other Pre Specified Outcome: Association of Biomarker With Overall Response Rate - P16 Status
Description: as for outcome 6
Time Frame: Up to 22 months
Population: Only the Head and Neck cancer cohort is being reported. No specimens were collected in the non-small cell lung cancer cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 0
Participants
  P16 Negative who achieved CR/PR: number analyzed (Participants) | 15 | 0
  P16 Negative who achieved CR/PR | 5 |
  P16 Positive who achieved CR/PR: number analyzed (Participants) | 10 | 0
  P16 Positive who achieved CR/PR | 1 |
Statistical Analysis 1: Comparison: Head and Neck Cancer Cohort; Test type: Other; p = 0.34, Fisher Exact

8. Other Pre Specified Outcome: Association of Biomarkers With Overall Response Rate - EphrinB2 Status
Description: as for outcome 6
Time Frame: Up to 22 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 0
Participants
  EphrinB2 Negative who achieved CR/PR: number analyzed (Participants) | 9 | 0
  EphrinB2 Negative who achieved CR/PR | 9 |
  EphrinB2 Positive who achieved CR/PR: number analyzed (Participants) | 16 | 0
  EphrinB2 Positive who achieved CR/PR | 6 |
Statistical Analysis 1: Comparison: Head and Neck Cancer Cohort; Test type: Other; p = 0.057, Fisher Exact

9. Other Pre Specified Outcome: Association of Biomarkers With Overall Response Rate - PD-L1 Status
Description: as for outcome 6
Time Frame: Up to 22 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 0
Participants
  PD-L1 Negative who achieved CR/PR: number analyzed (Participants) | 13 | 0
  PD-L1 Negative who achieved CR/PR | 3 |
  PD-L1 Positive who achieved CR/PR: number analyzed (Participants) | 12 | 0
  PD-L1 Positive who achieved CR/PR | 3 |
Statistical Analysis 1: Comparison: Head and Neck Cancer Cohort; Test type: Other; p = 1.00, Fisher Exact

10. Other Pre Specified Outcome: Association of Biomarkers With Overall Response Rate - EphrinB2 Positive/HPV-negative
Description: as for outcome 6
Time Frame: Up to 22 months
Population: Only the Head and Neck cancer cohort is being reported. No statistical analysis performed. No specimens were collected in the non-small cell lung cancer cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 11 | 0
Participants | 5 |

11. Other Pre Specified Outcome: Association of Biomarkers With Overall Survival (OS) - HPV Status
Description: OS was calculated from study entry to date of death. Participants last known to be alive are censored at date of last contact.
Time Frame: Up to 34 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 0
Months
  HPV Negative: number analyzed (Participants) | 15 | 0
  HPV Negative | 8.6 [2.0 to 12.6] |
  HPV Positive: number analyzed (Participants) | 10 | 0
  HPV Positive | 7.0 [1.5 to 28.8] |
Statistical Analysis 1: Comparison: Head and Neck Cancer Cohort; Test type: Other; p = 0.83, Log Rank

12. Other Pre Specified Outcome: Association of Biomarkers With Overall Survival (OS) - P16 Status
Description: as for outcome 11
Time Frame: Up to 34 months
Population: Only the Head and Neck cancer cohort is being reported. 10 participants were P16-positive, 15 participants were P16-negative, for a total of 25 participants. No specimens were collected in the non-small cell lung cancer cohort.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 0
Months
  P16 Negative: number analyzed (Participants) | 15 | 0
  P16 Negative | 8.6 [2.0 to 12.6] |
  P16 Positive: number analyzed (Participants) | 10 | 0
  P16 Positive | 7.0 [1.5 to 28.8] |
Statistical Analysis 1: Comparison: Head and Neck Cancer Cohort; Test type: Other; p = 0.83, Log Rank

13. Other Pre Specified Outcome: Association of Biomarkers With Overall Survival (OS) - EphrinB2
Description: as for outcome 11
Time Frame: Up to 24 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 0
Months
  EphrinB2 Negative: number analyzed (Participants) | 9 | 0
  EphrinB2 Negative | 7.0 [0.3 to 14.4] |
  EphrinB2 Positive: number analyzed (Participants) | 16 | 0
  EphrinB2 Positive | 10.9 [3.2 to 22.8] |
Statistical Analysis 1: Comparison: Head and Neck Cancer Cohort; Test type: Other; p = 0.83, Log Rank

14. Other Pre Specified Outcome: Association of Biomarkers With Overall Survival (OS) - PD-L1 Status
Description: as for outcome 11
Time Frame: Up to 34 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 0
Months
  PD-L1 Negative: number analyzed (Participants) | 13 | 0
  PD-L1 Negative | 12.3 [2.8 to 34.0] |
  PD-L1 Positive: number analyzed (Participants) | 12 | 0
  PD-L1 Positive | 7.6 [2.0 to 22.8] |
Statistical Analysis 1: Comparison: Head and Neck Cancer Cohort; Test type: Other; p = 0.47, Log Rank

15. Other Pre Specified Outcome: Association of Biomarkers With Overall Survival (OS) - EphrinB2 Positive/HPV-negative
Description: as for outcome 11
Time Frame: Up to 34 months
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 11 | 0
Months | 10.9 [2.0 to 13.7] |

16. Other Pre Specified Outcome: Association of Biomarkers With Progression Free Survival (PFS) - HPV Status
Description: From study entry to the date of first documented disease progression or death due to any cause, whichever came first.
Time Frame: Up to 11 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 0
Months
  HPV Negative: number analyzed (Participants) | 15 | 0
  HPV Negative | 2.5 [1.1 to 5.4] |
  HPV Positive: number analyzed (Participants) | 10 | 0
  HPV Positive | 2.6 [1.3 to 4.1] |
Statistical Analysis 1: Comparison: Head and Neck Cancer Cohort; Test type: Other; p = 0.83, Log Rank

17. Other Pre Specified Outcome: Association of Biomarkers With Progression Free Survival (PFS) - P16 Status
Description: From study entry to the date of first documented disease progression or death due to any cause, whichever came first.
Time Frame: Up to 11 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 0
Months
  P16 Negative: number analyzed (Participants) | 15 | 0
  P16 Negative | 2.5 [1.1 to 5.4] |
  P16 Positive: number analyzed (Participants) | 10 | 0
  P16 Positive | 2.6 [1.3 to 4.1] |
Statistical Analysis 1: Comparison: Head and Neck Cancer Cohort; Test type: Other; p = 0.83, Log Rank

18. Other Pre Specified Outcome: Association of Biomarkers With Progression Free Survival (PFS) - EphrinB2 Status
Description: From study entry to the date of first documented disease progression or death due to any cause, whichever came first.
Time Frame: Up to 11 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 0
Months
  EphrinB2 Negative: number analyzed (Participants) | 9 | 0
  EphrinB2 Negative | 2.5 [0.3 to 4.0] |
  EphrinB2 Positive: number analyzed (Participants) | 16 | 0
  EphrinB2 Positive | 2.9 [1.3 to 6.0] |
Statistical Analysis 1: Comparison: Head and Neck Cancer Cohort; Test type: Other; p = 0.11, Log Rank

19. Other Pre Specified Outcome: Association of Biomarkers With Progression Free Survival (PFS) - PD-L1 Status
Description: From study entry to the date of first documented disease progression or death due to any cause, whichever came first.
Time Frame: Up to 11 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 25 | 0
Months
  PD-L1 Negative: number analyzed (Participants) | 13 | 0
  PD-L1 Negative | 2.8 [1.2 to 5.6] |
  PD-L1 Positive: number analyzed (Participants) | 12 | 0
  PD-L1 Positive | 2.5 [1.2 to 5.4] |
Statistical Analysis 1: Comparison: Head and Neck Cancer Cohort; Test type: Other; p = 0.96, Log Rank

20. Other Pre Specified Outcome: Association of Biomarkers With Progression Free Survival (PFS) - EphrinB2 Positive/HPV-negative
Description: From study entry to the date of first documented disease progression or death due to any cause, whichever came first.
Time Frame: Up to 11 months
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 11 | 0
Months | 3.2 [1.1 to 7.3] |

ADVERSE EVENTS:
Time Frame: Up to 41 months
Arm/Group | Head and Neck Cancer Cohort | Non-Small Cell Lung Cancer Cohort
All-Cause Mortality (participants affected / at risk) | 12/25 | 6/17
Serious Adverse Events (participants affected / at risk) | 12/25 | 8/17
Other Adverse Events (participants affected / at risk) | 16/25 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Head and Neck Cancer Cohort (N=25) | Non-Small Cell Lung Cancer Cohort (N=17)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Alkaline Phosphatase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 2 | 0
Blood Bilirubin Increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypertension (Vascular disorders) | 9 | 6
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Colonic Perforation (Gastrointestinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pericolonic Abscess (Gastrointestinal disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Head and Neck Cancer Cohort (N=25) | Non-Small Cell Lung Cancer Cohort (N=17)
Hypertension (Vascular disorders) | 7 | 5
Fatigue (General disorders) | 3 | 5
Alanine Aminotransferase Increased (Investigations) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Weight loss (Investigations) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2
Alkaline Phosphatase Increased (Investigations) | 0 | 1
Creatinine Increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT03049618/Prot_SAP_000.pdf